CLINICAL TRIAL: NCT00873938
Title: Compliance to Artesunate-Amodiaquine Therapy for Uncomplicated Malaria in Rural Ghana
Acronym: Compliance
Status: Completed | Type: Observational
Sponsor: Kintampo Health Research Centre, Ghana (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Kwaku Poku Asante, Kintampo Health Research Centre
Other Study IDs: 2004/GD/70
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Malaria
Keywords: Artesunate-Amodiaquine; Compliance; Malaria
MeSH Terms: conditions — Malaria; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1-supervised
- 2 -unsupervised

SUMMARY:
With a change in malaria treatment policy to use combination antimalaria therapy, it is envisaged that compliance to combination therapy would be less than that of monotherapy that was being used for case management in Ghana. This is especially so as amodiaquine is unpopular because of its side-effects and the combination therapy is not a single formulation (fixed dose). Compliance may further be enhanced by community supervision through home visits of combination antimalarial therapy in cases of uncomplicated malaria.

This study would assess compliance to Artesunate-Amodiaquine therapy. It would also assess the effect of compliance to artesunate-amodiaquine therapy on clinical and parasitological cure rates. This study targeting age groups above ten years, would complement a child artesunate -amodiaquine efficacy study being undertaken by the same investigators in children ten years and below at Kintampo District at the same time. The funding for the child study has been approved by the Gates Malaria Partnership. Findings from both studies, involving all age groups would be made available to the National Malaria Control Programme and other stakeholders as practical information that may be beneficial to implementing policy change process from antimalarial monotherapy to a combination therapy.

DETAILED DESCRIPTION:
Primary objective:

• To determine compliance to artesunate-amodiaquine therapy among patients diagnosed with acute uncomplicated malaria in the Kintampo District Hospital.

Secondary objectives:

1. To determine patients compliance to each of the two drugs (artesunate or amodiaquine )
2. To determine reasons for differential compliance to either of the two drugs (artesunate or amodiaquine).
3. To determine patients perception and acceptance of artesunate-amodiaquine therapy for acute uncomplicated malaria.
4. To determine the effect of compliance of artesunate-amodiaquine therapy on clinical and parasitological improvement in acute uncomplicated malaria.

Study design: The study will be a pragmatic randomized control trial. Patients will be recruited based on an inclusion criteria stated below. Baseline clinical symptoms of malaria and presence of malaria parasite (Plasmodium falciparum) in the blood of eligible patients reporting sick at the health facility would be determined. Study patients would be randomized into one of two groups, intervention and control groups.

Intervention:

The intervention refers to supervisory home visits by a trained community volunteer to ensure that paticipants comply to treatment during the artesunate-amodiaquine therapy. Supervisory home visits by a trained community volunteer form a major component of the Community Health Planning and Services programme being implemented by the Ghana Health Service. The intervention group would be supervised during artesunate-amodiaquine therapy and the control group would not be supervised during artesunate-amodiaquine therapy. The primary and secondary outcome measures below will be determined and compared among the intervention and control group

Primary outcome measure:

The main outcome is compliance to artesunate-amodiaquine combination therapy. It is defined as no artesunate or amodiaquine left on the fourth day after start of treatment of a malaria episode. This would be assessed by the investigators direct observation of the blister package of artesunate-Amodiaquine tablets.

Secondary outcome measures:

* Reasons for non-compliance would be determined by response of study participants. Care-takers of children below 18 years will answer on behalf of their children with the child's assent.
* Participants' perception and acceptance of supervision: It would be assessed by responses given by study participants in an indepth interview.
* Parasite clearance rates on day 14 and 28 i.e. the proportion of study participants in each group with P. falciparum parasiteamia at day 14 and 28 determined by blood smear microscopy.
* Clinical cure rates by days 14 and 28 i.e. the proportion of study participants in each group with symptoms of malaria on days 14 and 28 determined by a structured questionnaire at these times.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients aged above ten years reporting at the Kintampo district hospital.
* Diagnosed as having Plasmodium falciparum uncomplicated malaria.
* Axillary temperature ≥37.5oC but less than 40 oC or history of fever in preceding 24 hr.
* Ability to tolerate oral therapy.
* Patient who live and can be located in the Kintampo District.
* Consent of patient and/or care giver (in the case of children)

Exclusion criteria:

* Pregnant women.
* Children ten years and below (to be catered for in the child antimalarial efficacy studies mentioned above).

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A rural population in the middle belt of Ghana
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The main outcome is compliance to artesunate-amodiaquine combination therapy | Within first three days after diagnosis of malaria

SECONDARY OUTCOMES:
Reasons for non-compliance | Within 28 days after diagnosis of malaria
Participants' perception and acceptance of supervision | Within 28 days after diagnosis of malaria
Parasite clearance rates on day 14 and 28 | Within 28 days after diagnosis of malaria

CONTACTS AND LOCATIONS:
Overall Officials: Seth Owusu-Agyei, PhD, Principal Investigator — Kintampo Health Research Centre, Ghana; Kwaku P Asante, MD, MPH, Principal Investigator — Kintampo Health Research Centre, Ghana
Locations (1):
- Kintampo Health Research Centre, Brong Ahafo Region, Kintampo, Ghana

REFERENCES:
- See also: Institutional Website, Kintampo Health Research Centre — http://www.kintampo-hrc.org/